CLINICAL TRIAL: NCT01593943
Title: Gender Equity-Focused, Male-Centered Family Planning for Rural India
Acronym: CHARM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Indian Council of Medical Research (Other Government); Population Council (Other)
Responsible Party: Principal Investigator, Anita Raj, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD061115 (NIH)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Family Planning
Keywords: contraception; india; rural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Condition (No Intervention)
- CHARM Intervention (Experimental): CHARM will be conducted via three 30-minute counseling sessions delivered in a rural setting, with the first session being required and the subsequent sessions being optional. The first two CHARM sessions will be for men only to build family planning (FP) and gender equity (GE) awareness and investment, and the third session will be for the couple with an emphasis on FP services, shared decision-making and marital communication. The three sessions can occur anytime within a 3 month timeframe but with a minimum of 1 week between sessions. All sessions and FP services (pill, condom, EC) will be provided at no cost to patients.
  Interventions: Behavioral: CHARM

INTERVENTIONS:
Behavioral: CHARM — CHARM will be conducted via three 30-minute counseling sessions delivered in the rural setting, with the first session required and the 2nd and 3rd sessions optional. The first two CHARM sessions will be for men only to build family planning (FP) and gender equity (GE) awareness and investment, and the third session will be for the couple with an emphasis on FP services, shared decision-making and marital communication. The three sessions can occur anytime within a 3 month timeframe but with a minimum of 1 week between sessions. All sessions and FP services (pill, condom, EC) will be provided at no cost to patients.
  Arms: CHARM Intervention

SUMMARY:
The major barrier to India meeting its national goal of replacement fertility is the huge discrepancy between urban and rural family planning, with rural young women at highest risk for unplanned and unspaced pregnancies. These concerns are considered to drive the persistent and unacceptably high rates of maternal and infant mortality in India. Major impediments to these young wives' acquisition of family planning services include high male partner control over reproductive decision-making, low mobility, and very low access to family planning services in villages. Such findings document the need for male-centered family planning efforts available at the village level, to better meet the needs of rural young wives. These male-centered efforts must address male gender role and gender inequity ideologies and norms (e.g., son preference, wife abuse) and marital communication, as these factors are associated with lower likelihood of contraceptive use in rural young Indian couples. Hence, the proposed study involves development and testing of the CHARM Program, a gender equity (GE)-focused, male-centered family planning (FP) program delivered by village health providers (VHPs), via a public-private partnership with primary health centers (PHCs) and private providers serving rural India. In Phase 1 the investigators will conduct formative research including health care resource mapping of Vasai within the Thane district of Maharashtra to identify villages and VHPs for inclusion in subsequent research and intervention. The investigators will also conduct in-depth interviews with rural young husbands (n=30), rural young wives (n=20), and health care providers (n=12), as well as focus groups with mothers' of rural young husbands (n=40). These data will be used to develop the CHARM program and efficacy trial. Phase 2 will involve development and pilot testing of CHARM protocols and training of VHPs for their role in the intervention trial (Phase 3). The CHARM intervention will involve VHP-delivered GE and FP counseling. It is delivered via a single session with 2 optional additional sessions one of which would include their wife. Phase 3 will involve evaluation of CHARM, using a two-armed randomized controlled trial design. Villages (N=50) will be randomized to receive either CHARM or the control program (standard FP referral to government public health centers [PHCs] located outside of villages), to assess treatment impact on spacing contraceptive use, pregnancy, and unmet family planning need. Intervention effects will be assessed via behavioral surveys with rural young husbands (18-30 years) and their wives (N=1000 couples, 20 couples per village) at baseline and 9 and 18 month follow-up, as well as pregnancy tests from wives, conducted at baseline and 18 month follow-up. A process evaluation will be undertaken via interviews with study participants and VHPs, as well as through VHP interviews and clinical record review, to assess program adherence, participation rates, response to program, and ease of delivery. In-depth interviews will also be conducted with key informants from the village and public and rural health systems to assess sustainability and institutionalization of the model.

ELIGIBILITY:
Primary study participants for intervention evaluation are rural young men (n=1500) and their wives (n=1500). Inclusion and exclusion criteria for these men are as follows:

INCLUSION CRITERIA

* Age 18-30 years and Fluent in Marathi
* Willing to Have Wife Included in the Study
* Residing in the village for the past 2 years and residing with wife in village for past 3 months

EXCLUSION CRITERIA

* Sterile or Wife is Sterile
* Cognitive Impairment (husband or wife)
* Intend to move in next 18 months

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2162 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
contraception | past 3 months
  female reports of contraceptive use (any and consistent) in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anita Raj, PhD, Principal Investigator — UCSD; Niranjan Saggurti, PhD, Principal Investigator — Population Council; Donta Balaiah, PhD, Principal Investigator — NIRRH
Locations (1):
- NIRRH, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Nair S, Dixit A, Ghule M, Battala M, Gajanan V, Dasgupta A, Begum S, Averbach S, Donta B, Silverman J, Saggurti N, Raj A. Health care providers' perspectives on delivering gender equity focused family planning program for young married couples in a cluster randomized controlled trial in rural Maharashtra, India. Gates Open Res. 2019 Jul 17;3:1508. doi: 10.12688/gatesopenres.13026.1. eCollection 2019. PMID 32266327
- [Derived] Shakya HB, Dasgupta A, Ghule M, Battala M, Saggurti N, Donta B, Nair S, Silverman J, Raj A. Spousal discordance on reports of contraceptive communication, contraceptive use, and ideal family size in rural India: a cross-sectional study. BMC Womens Health. 2018 Sep 4;18(1):147. doi: 10.1186/s12905-018-0636-7. PMID 30180845
- [Derived] Raj A, Ghule M, Ritter J, Battala M, Gajanan V, Nair S, Dasgupta A, Silverman JG, Balaiah D, Saggurti N. Cluster Randomized Controlled Trial Evaluation of a Gender Equity and Family Planning Intervention for Married Men and Couples in Rural India. PLoS One. 2016 May 11;11(5):e0153190. doi: 10.1371/journal.pone.0153190. eCollection 2016. PMID 27167981
- [Derived] Yore J, Dasgupta A, Ghule M, Battala M, Nair S, Silverman J, Saggurti N, Balaiah D, Raj A. CHARM, a gender equity and family planning intervention for men and couples in rural India: protocol for the cluster randomized controlled trial evaluation. Reprod Health. 2016 Feb 20;13:14. doi: 10.1186/s12978-016-0122-3. PMID 26897656